CLINICAL TRIAL: NCT00841529
Title: Evaluation of the Cardioblate Closure Device in Facilitating Occlusion of the Left Atrial Appendage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Medtronic Business Decision
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D02940
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Left Atrial Appendage Occlusion
Keywords: left atrial appendage; LAA; atrial fibrillation; AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Medtronic LAA Occlusion Device — Placement of the occlusion band on the LAA
  Other Names: Medtronic Cardioblate Closure Left Atrial Appendage Occlusion Device

SUMMARY:
The purpose of this study is to evaluate the performance of the Cardioblate Closure Device to occlude the LAA

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 18 years of age and less than or equal to 80 years of age
* Concomitant indication for cardiac surgery for one or more of the following:mitral valve repair or replacement, aortic valve repair or replacement, tricuspid valve repair or replacement, CABG (>=60 years of age), CABG (< 60 years of age with a history of atrial fibrillation), surgical ablation or Maze procedure
* The subject is willing and able to provide written informed consent and comply with study requirements
* The subject is not contra-indicated for intra-operative transesophageal echocardiogram (TEE)

Exclusion Criteria:

* Thrombus in the LAA and/or left atrium
* Prior LAA isolation attempts
* Subject is unable to take an anticoagulant during the study follow-up period
* Subject is undergoing an emergency cardiac procedure
* Life expectancy of less than 12 months
* Pregnancy or desire to be pregnant within the 12 months of the study procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Complete occlusion of the left atrial appendage | 3 Months

SECONDARY OUTCOMES:
To evaluate the composite incidence rate of device-related adverse events | Discharge/30 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCarthy, MD, Study Chair — Northwestern University
Locations (5):
- United States (5):
  - Eisenhower Medical Center, Rancho Mirage, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin